CLINICAL TRIAL: NCT06850753
Title: Superior Right Abdominal Excentration and Liver Transplantation (SURE-LT) for Perihilar Cholangiocarcinoma
Brief Title: En Bloc Resection of the Liver and Pancreas With a "Non-touch" Technique Followed by Liver Transplantation to Improve the Overall Survival in Patients With Non-resectable Hilar Cholangiocarcinoma Beyond the Mayo Clinic Transplant Criteria
Acronym: SURE-LT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Pål-Dag Line, Professor, Senior Consultant Transplant Surgeon, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK743190
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-02

CONDITIONS: Cholangiocarcinoma Non-resectable; Cholangiocarcinoma Recurrent; Liver Transplantation
Keywords: hilar cholangiocarcinoma; Liver transplantation
MeSH Terms: conditions — Klatskin Tumor | interventions — Pancreatic Hormones

STUDY DESIGN:
Intervention Model Description: Controlled prospective open-label trial to study liver transplantation in locally advanced hilar cholangiocarcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liver transplantation for locally advaced hilar cholangiocarcinoma (Experimental): Patients with hilar cholangiocarcinoma outside current transplant criteria will be treated with neoadjuvant chemotherapy + radiation and, after an observation period of a minimum of 6 months, undergo an exenteration of the liver and pancreas "en-bloc" + liver transplantation.
  Interventions: Procedure: Liver transplantation after en bloc resection of the liver and pancreas

INTERVENTIONS:
Procedure: Liver transplantation after en bloc resection of the liver and pancreas — Exenteration of the upper right part of the abdomen, including the liver and pancreas en bloc in locally advanced hilar cholangiocarcinoma, followed by liver transplantation

SUMMARY:
Surgery for hilar cholangiocarcinoma (phCCA) remains a significant challenge. The minority of patients who are eligible for resection are exposed to high procedure-related morbidity and mortality, and despite apparent R0 resection, cancer recurrence is common. The benefit of R1 resection compared to the best palliative chemotherapy has been questioned. The concept of extended surgery to achieve better radicality is controversial and in many instances, associated with higher procedure-related risk and unclarified oncological benefit. For unresectable patients, liver transplantation, per the Mayo protocol, remains the only alternative for a few patients.

Optimal staging pre- and intraoperatively is problematic since only the local biliary ductal involvement and, to a certain extent, lymph node dissemination can be reasonably correctly assessed. The reliability and validity of the intraoperative frozen section have been questioned. Furthermore, microscopic tumor cell affection leading to recurrent disease has been found in 16% of presumed N0 lymph nodes when analyzed by immunohistochemistry, and patients with nodal micrometastasis showed the same dismal survival as those with positive nodes on regular pathology (pN1).

Taken together, there is a lack of good surgical options for patients with marginally or unresectable phCCA that do not satisfy current criteria for liver transplantation.

The practical problem in the current surgical techniques for hilar cholangiocarcinoma, particularly in locally advanced disease, is that the hepatoduodenal ligament, in most instances, represents an incompletely staged operative field, making the probability of obtaining true free margins uncertain.

An alternative procedure must, therefore, consider the anatomical and multidimensional pattern of dissemination and the limitations in the accurate staging of phCCA, and this suggests that a wider surgical margin is needed to obtain radical resection in locally advanced phCCA.

The aim of the current study is tho these the following hypothesis:

Locally advanced hilar cholangiocarcinoma without M1 lymph node metastatic disease can be radically resected by extending the surgical margin to include the complete hepatobiliary axis and the main anatomical trajectories of local and regional dissemination through an "en-bloc" surgical approach.

M1 metastatic disease is defined as positive nodes in the following locations at staging:

* Station 9: lymph nodes around the celiac axis.
* Station 14: lymph nodes along the superior mesenteric artery or vein.
* Station 15: lymph nodes along the middle colic vein.
* Station 16: para-aortic lymph nodes.

Patients will be treated by chemotherapy and radiation therapy with an observation period of at least 6 months showing response or stable disease before final inclusion.

The operative procedure consists of a superior right abdominal exenteration, including the liver, pancreas, spleen, and vena cava + liver transplantation. If islets are available from the same donor, this will be administered postoperatively according to the institutional protocol.

Main enpoint is overall survival at 1, 3 and 5 years

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified or strong suspicion of cholangiocarcinoma based on radiology and endoscopy and elevated Ca 19-9 > 100U/L
* Perihilar cholangiocarcinoma that is deemed unresectable based on tumor location or severity of the underlying liver disease. Perihilar recurrence in PSC patients more than 24 months following the previous resection (N0, R0, no macrovascular involvement) is accepted.
* Patients should not be eligible for liver transplantation according to the Mayo protocol criteria.
* Tumor involvement of the hepatic artery distal to the gastroduodenal artery or the portal vein without tumor thrombus is accepted.
* No evidence of distant metastasis or metastatic lymph node (M1) involvement (para-aortic, coeliac or para-colic)
* Good performance status Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1
* At least 6 months of observation time during which the patient should be treated by chemotherapy and radiation (hyperfractioned 30-50 Gy) with response or stable disease before listing for LT. Patients with PSC and significant liver dysfunction that restricts the tolerability of chemoradiotherapy may be considered on an individual basis

Exclusion Criteria:

* Radiological signs of tumor invasion along intended resection borders
* Direct tumor invasion of the pancreatic head
* Signs of spread to the para-aortic, superior mesenteric, or coeliac lymph nodes
* Perforation of the visceral peritoneum
* Weight loss >10% in the last six months
* Patient BMI > 30 kg/m2
* Other malignancies, except curatively treated basal cell carcinoma or other tumors with disease-free interval > five years without relapse. The final decision on acceptable previous cancer diagnoses is at the principal investigator's discretion.
* Known history of human immunodeficiency virus (HIV) infection
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known hypersensitivity to rapamycin
* Prior metastatic disease
* Women who are pregnant or breastfeeding
* Any reason why, in the opinion of the investigator, the patient should not participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1, 3 and 5 years postoperatively
  Proportion of patients alive

SECONDARY OUTCOMES:
Disease-free survival | 1,3 and 5 years postoperatively
  Proportion of patients without evidence of disease
Survival after recurrence | months
  Survival time after diagnosis of cancer recurrence
Quality of life score | 6 and 12 months
  Quality of life will be measured using the European Organisation For Research And Treatment Of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30).
  The 30-item list captures key symptoms and signs related to bodily and mental function, and each item is scored on a scale of 1-4. The minimum score is 30, and the maximum is 120. A high score signifies a reduced quality of life.
Surgical complications | 90 days and 12 months
  Surgical complications according to the Clavien Dindo classification and the Comprehensive Complication Index.

CONTACTS AND LOCATIONS:
Overall Officials: Pål-Dag Line, MD PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
This is, for the time being, a single-site study. If the study is to include one or more sites, the IPD information will be shared.